CLINICAL TRIAL: NCT01453829
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Into the Internal Carotid Artery and Intravenously in Patients After Stroke
Brief Title: Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells in Patients After Stroke
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no enrolled participants
Sponsor: Ageless Regenerative Institute (Industry)
Collaborators: Instituto de Medicina Regenerativa (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-ST-ME-001
Record Dates: First submitted 2011-10-03; First posted 2011-10-18 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Harvesting and Isolation of Stem Cells — This will be an open-label, non-randomized multi-center patient sponsored study of ASC implantation using a catheter delivery system. ASCs will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The cells will be implanted into the Internal Carotid Artery and intravenously.

SUMMARY:
The intent of this clinical study is to answer the questions:

1. Is the proposed treatment safe
2. Is treatment effective in improving the disease pathology of patients after Stroke and clinical outcomes?

DETAILED DESCRIPTION:
Adipose-Derived Stromal Cells (ASCs) are a novel therapy for patients suffering from stroke. By injecting ASCs either into the internal carotid artery, these regions may become populated with the ASCs, thereby potentially restoring brain function. ASCs are a patient-derived ("autologous") cell transplantation technology that is delivered to the patient into the internal carotid artery and intravenously. The therapy is composed of cells derived from a patients' own adipose tissue that are isolated within approximately 1 hour and immediately delivered back to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 18 and 80 years.
* Symptoms and signs of clinically definite ischemic stroke or hemorrhagic stroke
* DWI-MRI has reliably shown relevant ischemic lesions
* Extracranial duplex/transcranial Doppler must confirm intra/extracranial arteries permeability
* The stroke is severe (NIH Stroke Scale >= 8 before procedure)
* Up to date on all age and gender appropriate cancer screening per American Cancer Society.

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease and/or known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis will have expert consultation to determine eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg or greater than 180mmHg
* Resting heart rate > 100 bpm;
* Active clinical infection being treated by antibiotics within one week of enrollment.
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in clinical function from baseline as assessed by the NIH stroke scale at three months | 3 months
Number of participants with adverse events | 1 week
  The safety of adipose-derived stem cell injection will be evaluated by assessment of the frequency and nature of adverse events occurring during the study injection and up to the 6-month period following treatment.
Number of participants with adverse events at 2 weeks | two weeks
Number of participants with adverse events at 4 weeks | 4 weeks
Improvement in clinical function from baseline as assessed by the NIH stroke at 6 months | 6 months
Number of participants with adverse events at 3 weeks | 3 weeks
Improvement in clinical function as assessed by Barthel Scale compared to baseline at 6 months | 6 months

SECONDARY OUTCOMES:
Improvement in clinical function as assessed by Modified Rankin Score compared to baseline at 3 months | 3 months
Improvement in clinical function as assessed by Barthel Scale compared to baseline at 3 months | 3 months
Improvement in Magnetic resonance imaging (MRI) scan compared to baseline at three months | 3 months
Improvement in clinical function as assessed by Modified Rankin Score compared to baseline at 6 months | 6 months
Improvement in clinical function as assessed by Barthel Scale compared to baseline at 6 months | 6 months
Improvement in Magnetic resonance imaging (MRI) scan compared to baseline at six months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Victor D Morales, MD, Principal Investigator — Instituto de Medicina Regenerativa; Clemente Zuñiga, MD, Principal Investigator — Instituto de Medicina Regenerativa
Locations (1):
- Hospital Angeles, Tijuana, Estado de Baja California, Mexico